CLINICAL TRIAL: NCT01026844
Title: A Phase I Study of Hydroxychloroquine With or Without Erlotinib in Advanced NSCLC
Brief Title: Hydroxychloroquine With or Without Erlotinib in Advanced Non-small Cell Lung Cancer (NSCLC)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: slow enrollment
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Lecia V. Sequist, PI, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07-037; OSI4251s (Other: Genentech)
Record Dates: First submitted 2009-12-02; First posted 2009-12-04 (Estimated); Results first posted 2013-07-31 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2017-01

CONDITIONS: Non-small Cell Lung Cancer
Keywords: erlotinib; tarceva; hydroxychloroquine; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride; Hydroxychloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Erlotinib plus hydroxychloroquine (Experimental): erltoinib 150mg per day plus HCQ in esclating doses of 400mg, 600mg, 800mg and 1000mg per day
  Interventions: Drug: erlotinib; Drug: hydroxychloroquine
- Hydroxychloroqine (Experimental): hydroxychloroquine given at escalating doses of 400mg, 600mg, 800mg and 1000mg per day
  Interventions: Drug: hydroxychloroquine

INTERVENTIONS:
Drug: erlotinib — Taken orally once a day
  Other Names: Tarceva
  Arms: Erlotinib plus hydroxychloroquine
Drug: hydroxychloroquine — Taken orally once a day
  Other Names: HCQ

SUMMARY:
Erlotinib is a type of drug called a tyrosine kinase inhibitor (TKI). TKIs block a protein called epidermal growth factor receptor (EGFR). EGFR may control tumor growth and tumor cell survival. EGFR is found on the surface of many types of cancer cells, including non-small cell lung cancer (NSCLC). Erlotinib is approved by the Food and Drug Administration (FDA) for the treatment of NSCLC. Hydroxychloroquine (HCQ) is a drug approved by the FDA for treatment of malaria, rheumatoid arthritis, and several other diseases but is not currently thought of as a cancer treatment. Previous laboratory studies suggests that HCQ may have an anti-cancer effect by itself in some situations, particularly when EGFR TKI drugs have been useful in the past against the tumor. The two drugs together may be able to fight lung cancer in cases where erlotinib is no longer effective by itself. The purpose of this research study is to determine the highest dose of HCQ that can be given safely in combination with erlotinib. We will also begin to look at whether HCQ plus erlotinib helps treat cancer that have become resistant to TKI treatment after initially responding.

DETAILED DESCRIPTION:
* The goal of this study is to find the highest dose of HCQ that can be given safely with erlotinib. Therefore, not all participants will receive the same dose of HCQ. Small groups of participants will be enrolled in steps in this trial. The first group will be given a certain dose of HCQ. If they have few or manageable side effects, the next small group of participants enrolled will receive a higher dose. This increase in doses will continue until the research doctors find the highest dose of HCQ that can be given without causing severe or unmanageable side effects.
* Both HCQ and erlotinib are pills that are taken orally. Treatment will be divided into time periods called cycles. Each treatment cycle is 28 days. The exception to this 28 day cycle is when participants start taking the pills for the first time. Erlotinib is started first for 7 days and then HCQ is added. When the HCQ begins, the first cycle of 28 days begins.
* There are several tests and procedures that will be performed at specific time periods during protocol treatment. These include: blood work, performance status assessment, questions about medical history and medications, tumor assessment with CT or MRI and, eye exams.
* Participants may continue to receive study treatment as long as they do not experience unacceptable side effects or disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed diagnosis of non-small cell lung cancer
* Stage IIIB with pleural effusion or Stage IV disease by the American Joint Committee on Cancer (AJCC) 6th edition staging criteria.
* At least 12 weeks of prior treatment with erlotinib, gefitinib, or another EGFR small molecule TKI agent.
* Age equal to or greater than 18 years
* Measurable disease, defined according to RECIST criteria
* Performance status of 0, 1 or 2
* At least 2 weeks since prior radiation treatment
* At least 2 weeks since any prior chemotherapy or targeted therapy
* Adequate organ function as outlined in the protocol
* Approval for HCQ treatment by an eye doctor, based on a screening eye exam. Examples of disqualifying baseline conditions include macular degeneration and other retinal disease.
* Willingness to comply with protocol procedures including the blood-sampling schedule for PK analyses and periodic eye examination

Exclusion Criteria:

* Current use of hydroxychloroquine for any reason
* Known hypersensitivity to chloroquine, hydroxychloroquine, or any other closely related drug
* Known hypersensitivity to erlotinib, gefitinib, or any closely related drug
* Glucose-6-phosphate dehydrogenase (G6PD) deficiency, as HCQ may cause hemolytic anemia in patients with G6PD deficiency
* Cataracts that would interfere with required funduscopic examinations, or severe baseline visual impairment including macular degeneration, retinopathy or visual field changes, or having only one functional eye. All patients must undergo a screening eye exam prior to enrollment
* Pregnancy or breastfeeding. Female subjects of childbearing age and male subjects must practice acceptable method of birth control
* Symptomatic CNS metastases or newly diagnosed CNS metastases that have not yet been definitively treated with radiation and/or surgery
* Prior radiation therapy inclusive of all identified target lesions
* Any evidence of clinically active interstitial lung disease
* Malignancies within the past 3 years except for adequately treated carcinoma of the cervix or basal or squamous cell carcinomas of the skin
* Although not an absolute exclusion criteria, caution should be exercised in patients with a diagnosis of porphyria or non-light sensitive psoriasis, as HCQ can significantly exacerbate both of those conditions
* Evidence of any other significant clinical disorder or laboratory finding that makes it undesirable for the patient to participate in the study
* Use of any non-FDA approved or investigational agent within 2 weeks of enrolling onto the trial, or failure to recover from the side effects of any of these agents
* Penicillamine use for Wilson's disease or any other indication, as concomitant use with HCQ can increase toxicity to penicillamine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2007-07; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lecia Sequist, MD, MPH, Principal Investigator — Massachussets General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Result] Goldberg SB, Supko JG, Neal JW, Muzikansky A, Digumarthy S, Fidias P, Temel JS, Heist RS, Shaw AT, McCarthy PO, Lynch TJ, Sharma S, Settleman JE, Sequist LV. A phase I study of erlotinib and hydroxychloroquine in advanced non-small-cell lung cancer. J Thorac Oncol. 2012 Oct;7(10):1602-8. doi: 10.1097/JTO.0b013e318262de4a. PMID 22878749

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twenty-seven patients were enrolled between August 2007 and May 2010. They were all patients at Mass General Hospital Cancer Center
Groups:
- Erlotinib Plus HCQ (Hydroxychloroquine): Erlotinib at 150mg QD and HCQ at escalating doses (400mg, 600mg, 800mg and 1000mg QD)
- HCQ (Hydroxychloroquine): HCQ at escalating doses (400mg, 600mg, 800mg, and 1000mg QD)
Period: Overall Study
Arm/Group | Erlotinib Plus HCQ (Hydroxychloroquine) | HCQ (Hydroxychloroquine)
Started | 19 | 8
Completed | 19 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Erlotinib Plus HCQ (Hydroxychloroquine) | HCQ (Hydroxychloroquine) | Total
Number analyzed (Participants) | 19 | 8 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 6 | 15
  >=65 years | 10 | 2 | 12
Age, Continuous [Median (Full Range); unit: years] | 65 [27 to 73] | 61 [48 to 76] | 64 [27 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 5 | 15
  Male | 9 | 3 | 12
Region of Enrollment [Number; unit: participants]
  United States | 19 | 8 | 27

OUTCOME MEASURES:

1. Primary Outcome: Describe the Number and Type of Observed Dose Limiting Toxcities
Description: HCQ doses tested included 400mg, 600mg, 800mg, and 1000mg. Dose-limiting toxicities (DLTs) were defined as CTC of grade 2 or higher retinopathy or keratitis, or CTC of grade 3 or higher hematologic, skin, CNS, neuropathic, cardiac, respiratory, gastrointestinal, or renal AEs in the first cycle considered at least possibly related to HCQ. If a DLT was observed, an additional three patients were enrolled at that dose level. The maximum tolerated dose for HCQ in each arm would be defined as one dose level below that at which two or more of 6 patients experienced a DLT, or if no DLTs were observed, the highest tested dose.
Time Frame: 2 years
Population: In October 2008, after enrollment of 18 patients (8 on arm A and 10 on arm B), the study was amended to limit enrollment to arm B only (HCQ plus erlotinib) given the increasing preclinical evidence supporting a role for combination therapy (but not HCQ monotherapy) and to help increase overall patient accrual.
Measure: Number; unit: participants
Arm/Group | Erlotinib Plus HCQ (Hydroxychloroquine) | HCQ (Hydroxychloroquine)
Number analyzed (Participants) | 19 | 8
participants | 0 | 0

2. Secondary Outcome: Determine the Pharmacokinetic (PK) Parameters of Hydroxychloroquine (HCQ) Plus Erlotinib.
Description: PK parameter tested was dose normalized minimum steady state concentration (Cmin SS) of HCQ in micromolar per gram. Note this outcome was only analyzed for the first 21 patients enrolled, 13 on erlotinib/HCQ and 8 on HCQ arm.
Time Frame: 2 years
Population: The patients participating in the randomized portion of the study were analyzed for PK parameters. When the HCQ alone arm of the study was closed, PK measurements were no longer performed
Measure: Mean (Standard Deviation); unit: micromolar per gram
Arm/Group | Erlotinib Plus HCQ (Hydroxychloroquine) | HCQ (Hydroxychloroquine)
Number analyzed (Participants) | 13 | 8
micromolar per gram | 5.93 (2.51) | 9.40 (5.85)

3. Secondary Outcome: Objective Tumor Response Rate
Description: Number of Response Evaluation Criteria in Solid Tumors (RECIST) responses divided by number of patients treated. Per RECIST version 1.0 complete response (CR) is defined as disappearance of all target lesions; Partial Response (PR) is defined as >=30% decrease in the sum of the longest diameter of target lesions. The objective tumor response rate is the CR + PR divided by the total number of patients
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Erlotinib Plus HCQ (Hydroxychloroquine) | HCQ (Hydroxychloroquine)
Number analyzed (Participants) | 19 | 8
percentage of patients | 5 [1 to 25] | 0 [0 to 34]

4. Secondary Outcome: Correlate Epidermal Growth Factor Receptor (EGFR) Mutations and EGFR Amplification With Response to Treatment in Patients With Available Tumor Specimens.
Time Frame: 2 years
Population: Because so few responses were observed, this exploratory outcome was not analyzed
Arm/Group | Erlotinib Plus HCQ (Hydroxychloroquine) | HCQ (Hydroxychloroquine)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Erlotinib Plus HCQ (Hydroxychloroquine) | HCQ (Hydroxychloroquine)
Serious Adverse Events (participants affected / at risk) | 6/19 | 0/8
Other Adverse Events (participants affected / at risk) | 15/19 | 4/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Erlotinib Plus HCQ (Hydroxychloroquine) (N=19) | HCQ (Hydroxychloroquine) (N=8)
rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
dehydration (Gastrointestinal disorders) | 1 (1) | 0 (0)
nail changes (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Erlotinib Plus HCQ (Hydroxychloroquine) (N=19) | HCQ (Hydroxychloroquine) (N=8)
rash (Skin and subcutaneous tissue disorders) | 10 (10) | 0 (0)
diarrhea (Gastrointestinal disorders) | 9 (9) | 0 (0)
nausea (Gastrointestinal disorders) | 9 (9) | 3 (3)
fatigue (General disorders) | 7 (7) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination of study leading to small numbers of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No